CLINICAL TRIAL: NCT04431206
Title: Generate a Pharmacodynamic Model of Oxytocin for Peripheral Analgesic Effects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data from the initial participants were analyzed to support an NIH grant submission, leading to NIH funding of a new protocol to expand on the initial results.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00066136
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee; Healthy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: All arms receive the same IV oxytocin 30-minute infusion. Participants are randomly assigned for heat pain testing every 15 min for 60 min beginning at either 2, 5, 7, or 10 minutes from the beginning of the IV oxytocin infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Verbal pain score at 2 minutes (Other): Verbal pain score is recorded at the end of 5 minutes of heating the skin. In this arm the first score is obtained at 2 minutes after starting the intervention, then every 15 minutes for 60 minutes
  Interventions: Drug: Oxytocin
- Verbal pain score at 5 minutes (Other): Verbal pain score is recorded at the end of 5 minutes of heating the skin. In this arm the first score is obtained at 5 minutes after starting the intervention, then every 15 minutes for 60 minutes
  Interventions: Drug: Oxytocin
- Verbal pain score at 7 minutes (Other): Verbal pain score is recorded at the end of 5 minutes of heating the skin. In this arm the first score is obtained at 7 minutes after starting the intervention, then every 15 minutes for 60 minutes
  Interventions: Drug: Oxytocin
- Verbal pain score at 10 minutes (Other): Verbal pain score is recorded at the end of 5 minutes of heating the skin. In this arm the first score is obtained at 10 minutes after starting the intervention, then every 15 minutes for 60 minutes
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 8.2 IU, administered by 30minute IV infusion starting at time 0
  Other Names: Pitocin

SUMMARY:
This is a study of participants that will receive an intravenous (IV) infusion of oxytocin (naturally occurring hormone that is made in the brain).

In this study healthy volunteers and people with knee arthritis so severe that they may need joint replacement are recruited for a one day study. Each study participant will have an IV catheter placed. After placement of the IV catheter oxytocin will be given by IV infusion. Investigators will perform some tests to evaluate how oxytocin changes perceptions on the skin. Investigators will study a painful perception by placing a probe on the skin and heating it to 113 -117 degrees Fahrenheit (F) for 5 minutes. Each study participant will score any pain that is experienced on a 0 to 10 scale, and most people find that pain rises during the 5 minutes, but remains mild, usually around only 1 or 2 on the 0 to 10 scale. The 5 minute heating temperature will be determined according to the subjects pain rating during the screening visit.

The main goal of the study is to determine the effect of oxytocin during and after a fixed rate intravenous infusion on reduction in pain to a sustained heat stimulus in order to generate a model for peripheral analgesia.

DETAILED DESCRIPTION:
In this study healthy people or those with knee arthritis so severe that they may need joint replacement are recruited for a one day study. Study participants will come to the Clinical Research Unit (CRU) and one intravenous (IV) catheter will be inserted in the forearm for oxytocin infusion. Participants in this study will receive oxytocin at a steady rate for 30 minutes. This information will be analyzed by another group at Stanford University in the Pharmacokinetic/Pharmacodynamic (PK/PD) Core part of this application. Mathematics will be utilized to calculate how quickly oxytocin moves from the blood to where it reduces pain.

Investigators will also do a pain test to determine how much oxytocin reduces pain. For this Investigators will place a probe on the skin and heat it to 113 - 117 degrees for 5 minutes. Study participants will score any pain they feel on a 0 to 10 scale, and most people find that pain rises during the 5 minutes, but remains mild, usually around only 1 or 2 on the 0 to 10 scale.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
5. Subjects with current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval.
6. Subjects with past or current history of hyponatremia or at risk for hyponatremia; anyone taking thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, Ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, SSRI's, MAOI, or the recreational drug ecstasy.
7. Subjects with a known latex allergy.
8. Subjects with a pain score rating of 1 or less during the initial training session to a 5 minute heating of 45°C- 47 °C to the lower calf.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be provided upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available upon posting results to a preprint server, anticipated to occur by the end of the first quarter of 2026
Access Criteria: For the purpose of pharmacokinetic / pharmacodynamic modeling or meta-analyses / review publications.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants were recruited from the community from October 15, 2020 through November 15, 2020 via IRB-approved advertisements and IRB-approved lists of previous participants who agreed to be contacted for future studies. They were recruited by phone and provided written informed consent at the day of the training visit.
Period: Overall Study
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
Started | 2 | 1 | 2 | 2
Completed | 2 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes | Total
Number analyzed (Participants) | 2 | 1 | 2 | 2 | 7
Age, Continuous [Mean (Full Range); unit: years] | 36 [32 to 40] | 34 [34 to 34] | 22.5 [22 to 23] | 25 [24 to 26] | 26 [22 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 3
  Male | 0 | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 2 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 0 | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 2 | 2 | 7
Verbal pain score at the end of 5 minute skin heating [Mean (Full Range); unit: units on a scale] | 3.0 [3.0 to 3.0] | 5.0 [5.0 to 5.0] | 3.5 [3.0 to 4.0] | 2.0 [2.0 to 2.0] | 3.1 [2.0 to 5.0]

OUTCOME MEASURES:

1. Primary Outcome: First Verbal Pain Score After Beginning IV Oxytocin Infusion
Description: Pain at the end of 5 minutes of heating the skin to 45 - 47 degrees C will be determined using a Verbal Pain scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to THE WORST PAIN IMAGINABLE. Heating temperature is determined by pain rating during screening visit.
Time Frame: 2-10 minutes after starting oxytocin infusion, depending on Arm
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
Number analyzed (Participants) | 2 | 1 | 2 | 2
units on a scale | 3.5 [3.0 to 4.0] | 4.0 [4.0 to 4.0] | 3.5 [3.0 to 4.0] | 1.5 [1.0 to 2.0]

2. Primary Outcome: Second Verbal Pain Score After Beginning IV Oxytocin Infusion
Description: as for outcome 1
Time Frame: 17-25 minutes after starting oxytocin infusion, depending on Arm
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
Number analyzed (Participants) | 2 | 1 | 2 | 2
units on a scale | 1.5 [1.0 to 2.0] | 3.0 [3.0 to 3.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0]

3. Primary Outcome: Third Verbal Pain Score After Beginning IV Oxytocin Infusion
Description: as for outcome 1
Time Frame: 32-40 minutes after starting oxytocin infusion, depending on Arm
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
Number analyzed (Participants) | 2 | 1 | 2 | 2
units on a scale | 3.0 [3.0 to 3.0] | 4.0 [4.0 to 4.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

4. Primary Outcome: Fourth Verbal Pain Score After Beginning IV Oxytocin Infusion
Description: as for outcome 1
Time Frame: 47-55 minutes after starting oxytocin infusion, depending on Arm
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
Number analyzed (Participants) | 2 | 1 | 2 | 2
units on a scale | 2.0 [1.0 to 3.0] | 3.0 [3.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]

5. Primary Outcome: Fifth Verbal Pain Score After Beginning IV Oxytocin Infusion
Description: as for outcome 1
Time Frame: 62-70 minutes after starting oxytocin infusion, depending on Arm
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
Number analyzed (Participants) | 2 | 1 | 2 | 2
units on a scale | 3.0 [3.0 to 3.0] | 2.0 [2.0 to 2.0] | 1.5 [1.0 to 2.0] | 0.5 [0.0 to 1.0]

ADVERSE EVENTS:
Time Frame: The oxytocin infusion day and the next 5 days
Description: Querying during and at intervals for any subjective sensations during and after oxytocin infusion on the study day. In addition, continuous recording of blood pressure, heart rate, and oxyhemoglobin saturation during oxytocin infusion and at regular intervals afterwards on the study day.
  Telephone calls daily with querying for any adverse events.
Arm/Group | Verbal Pain Score at 2 Minutes | Verbal Pain Score at 5 Minutes | Verbal Pain Score at 7 Minutes | Verbal Pain Score at 10 Minutes
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
The study was paused after the completion of 7 healthy participants and data were analyzed for the purpose of a grant application revision. The results led to a heavily revised proposed study of pharmacodynamic modeling, and when the grant was funded, this new study was approved and performed under a different IRB approval and CTG registration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04431206/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT04431206/ICF_001.pdf